CLINICAL TRIAL: NCT04746755
Title: An Open-label, Single-centre, Parallel-group Clinical Investigation, to Evaluate the Effectiveness and In-use Tolerability of a Range of Four Orthotic Insoles on Target Areas of Pain in the Lower Body, Associated With Musculoskeletal Stress, Experienced by Those Who Spend Most of Their Working Day on Their Feet
Brief Title: Effectiveness of Four Orthotic Insoles on Pain in the Lower Body Associated With Musculoskeletal Stress
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants experienced data collection issues when using the eDiary, these issues increased the burden and lowered compliance. Updates to the eDiary were unsuccessful at resolving the issues so the decision was taken to terminate the Investigation.
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: SynteractHCR Deutschland GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPD85302
Record Dates: First submitted 2021-01-29; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: An open-label, single-centre, parallel-group clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Lower back pain associated with musculoskeletal stress (Experimental): Subjects eligible for the study self selected the insole for the pain in-accordance with the pain that they were experiencing due to musculoskeletal stress. Subjects within this arm of the study experienced lower back pain; the subjects selection was corroborated by a physiotherapist.
  Interventions: Device: Orthotic Insole: Lower Back
- Experimental: Heel pain associated with musculoskeletal stress (Experimental): Subjects eligible for the study self selected the insole for the pain in-accordance with the pain that they were experiencing due to musculoskeletal stress. Subjects within this arm of the study experienced pain in the heels of their feet; the subjects selection was corroborated by a physiotherapist.
  Interventions: Device: Orthotic Insole: Heel
- Experimental: Knee to Heel pain associated with musculoskeletal stress (Experimental): Subjects eligible for the study self selected the insole for the pain in-accordance with the pain that they were experiencing due to musculoskeletal stress. Subjects within this arm of the study experienced Knee to Heel pain; the subjects selection was corroborated by a physiotherapist.
  Interventions: Device: Orthotic Insole: Knee to Heel
- Experimental: Arch pain associated with musculoskeletal stress (Experimental): Subjects eligible for the study self selected the insole for the pain in-accordance with the pain that they were experiencing due to musculoskeletal stress. Subjects within this arm of the study experienced pain in the arch of their feet; the subjects selection was corroborated by a physiotherapist.
  Interventions: Device: Orthotic Insole: Arch

INTERVENTIONS:
Device: Orthotic Insole: Lower Back — This Insole is a full-length shaped orthotic insole, with a heel cup and an arch support. The insole can cover several shoe sizes and can be cut to the correct size to fit in the shoe.
  Arms: Experimental: Lower back pain associated with musculoskeletal stress
Device: Orthotic Insole: Heel — This Insole is a horseshoe shaped flexible heel cup with a softer area where the heel would be expected.
  Arms: Experimental: Heel pain associated with musculoskeletal stress
Device: Orthotic Insole: Knee to Heel — This Insole is a ¾ length rigid orthotic insole with a softer area where the heel would be expected. Each insole will cover several shoe sizes.
  Arms: Experimental: Knee to Heel pain associated with musculoskeletal stress
Device: Orthotic Insole: Arch — This Insole is a ¾ length shaped medical device with a softer area incorporated into the ball of foot and heel area and an external arch.
  support and 6-8 mm metatarsal dome. The slim fit insole runs from the heel along under the arch of the foot and reaches to just behind the toes to prevent squashing the toes in tight fitting shoes.
  Arms: Experimental: Arch pain associated with musculoskeletal stress

SUMMARY:
This was an open-label, single-centre, parallel-group clinical investigation, to evaluate the effectiveness and in-use tolerability of a range of four orthotic insoles on target areas of pain in the lower body, associated with musculoskeletal stress, experienced by those who spend most of their working day on their feet

DETAILED DESCRIPTION:
This was an open-label, single-centre, parallel-group clinical investigation, to evaluate the effectiveness and in-use tolerability of a range of four orthotic insoles on target areas of pain in the lower body, associated with musculoskeletal stress, experienced by those who spend most of their working day on their feet.

The investigation design included two periods; 'run-in' period and 'treatment' period. The treatment period comprised of two sub-periods; a 'breaking-in' period and the 'full use' period. The breaking-in period was intended to allow time for the subjects' feet to accustom to wearing the insoles. The full-use period was used to determine effectiveness of the insoles. These periods constitute lengths of time defined for the purpose of the investigation as "working episodes". Working episodes were defined as at least 3 (up to 6) consecutive working days of at least 6 hours each at work, following at least 2 consecutive non-working days.

Eligible subjects at Visit 1 (screening) were enrolled into the run-in period, where subjects were assessed prior to treatment with the insoles under investigation. During the run-in period, consisting of one working episode, subjects self-reported their pain without using insoles on a daily basis (Q3-9 of the Brief Pain Inventory (BPI)), in order to provide the baseline data to which the insoles were compared. Eligible subjects were enrolled into the treatment period at Visit 2 and assigned the insole relevant to the target pain area/pain area combination. Insole use was built up gradually during a breaking-in period, which constituted one working episode, with at least one nonworking day prior to the start of the working episode. Following the breaking-in period, the full-use period commenced. During the treatment period, subjects wore the insoles on working days and as much as possible on non-working days, self-reporting their pain daily (BPI Questions 3 - 9 inclusive).

ELIGIBILITY:
Inclusion Criteria:

1. Those who gave informed consent.
2. Those who understood the purpose of the investigation, cooperate with the investigation procedures and tasks and were to attend the investigational site for all investigation assessments.
3. Those were willing to continue with their normal daily activities, including any cosmetic foot care regimens (including the use of products) throughout the investigation and not partake in exercise which is not normal for them and which would be deemed by the Investigator to impact study assessments, or any new foot care or podiatric treatments unless agreed in advance with the Investigator.
4. Those who wore the same or similar type of standard shoe during their working day/shift for at least the 4 weeks prior to enrolment (Visit 1) (or they have worn a different shoe which cause no change to their pain) and who were able to wear the same standard* shoe during their working day / shift for the duration of the investigation.

   Eligibility regarding this criterion was confirmed at Visit 1 but will also confirmed by the physiotherapist at Visit 2, following their assessment.

   *A standard shoe was defined as closed shoe, ≤2-inch heel, with an adequate sole, upper and toe box to accommodate the orthotic insole, as determined by the physiotherapist. Shoes with orthotic-type internal contouring (as determined by the physiotherapist to include features which could alter gait) or shoes with an arch support greater than 12 mm would not be permitted. Odour-eaters cannot be used during the treatment period.
5. Male and female subjects from the age of 18 years and a BMI of 18.5-29.9 kg/m² inclusive.
6. Those who had access to a mobile device (iOS or Android smart phone or tablet), with access to the internet, and are able to operate an app.
7. Those with a shoe size between 4.5 to 11 (UK).
8. Those who worked at least 30 hours per week which usually involved "working episodes"

   (defined as at least 3 (up to 6) consecutive working days (of at least 6 hours each at work) following at least 2 consecutive non-working days), which were expected to continue throughout their involvement in the investigation, and included at least 4 working episodes during the 4 (up to 5)-week treatment period.

   These working episodes should be non-complex in the opinion of the Investigator, to ensure continued eligibility.
9. Those who spent most (at least three quarters) of their working day on their feet, and remained in their current employment/work environment throughout the investigation period.
10. Those who have experienced pain associated with musculoskeletal stress during working episodes, for at least 4 weeks prior to enrolment (Visit 1) that they can distinguish as being in one of the following primary areas of pain or combination thereof, that the Investigator or designee considers could be treated with the relevant insole to be used in the investigation:

    * Lower back
    * Knee and/or Heel
    * Arch
    * Heel

    Eligibility regarding this criterion will also be confirmed by the physiotherapist at Visit 2, following their assessment.
11. Those who scored an average of 5 (±1) on the BPI average pain item (question 5) over the first three consecutive working days of the run-in period working episode**, when assessed specifically in their primary target pain area/pain area combination, as confirmed at Visit 2.

    * If the run-in period constituted more than one working episode (e.g. due to the scheduling of Visit 2), only the data from the first working episode was included in the calculation to determine eligibility, providing this included at least three consecutive working days. Otherwise data from the second working episode was used.

Exclusion Criteria:

1. Those who had a current medical condition that is contraindicated by the use of the orthotic insoles (e.g. peripheral vascular disease, sensory neuropathy or diabetes).
2. Those who currently use prescribed orthotics for biomechanical or other issues, or have received and used prescribed orthotics within the last 12 months or over-the-counter (OTC) orthotics in the last 6 months (odour-eaters and any non-structured/non-orthotic shock-absorber insole were permitted).
3. Those with any significant medical history which in the opinion of the Investigator could have interfered with the assessments of the investigation. For example; structural conditions (e.g. bunion or bunionette), lower limb or foot injury, rheumatic disease (e.g. rheumatoid arthritis, scleroderma, polymyalgia rheumatica), fibromyalgia, neurological disease or moderate to severe depression.
4. Those who were taking any of the following medications:

   1. Anti-psychotic, sedatives, muscle-relaxants or medicines intended to treat neuropathic pain
   2. Anti-inflammatory medications which would reduce systemic inflammation or locally at the target pain areas (low dose Aspirin (75 mg daily) and nasal/inhaled steroids could have been considered acceptable, where in the opinion of the Investigator they would not interfere with the assessments of the investigation)
   3. An unstable dose of anti-depressants (defined as a change in therapy within the last 6 months).
5. Those who are taking regular medication for targeted pain (including OTC pain relief, in excess of 2g paracetamol daily) which is either beyond the maximum recommended daily dose according to the SmPC or which the Investigator deems inappropriate for the subject to continue at the same dose throughout the investigation.
6. Those who were pregnant or who had given birth within the past 6 months.
7. Females of child-bearing potential who were unwilling to use a minimum of an "acceptable" (as defined by the Clinical Trials Facilitation Group (CFTG; 2014) recommendations) level of birth control, for the entire duration of the investigation.

   Suitable methods of birth control (in accordance with "highly effective" and "acceptable" methods of birth control defined by the CTFG) included:
   1. Combined (estrogen and progestogen containing) hormonal contraception associated with the inhibition of ovulation; oral, intravaginal, transdermal.
   2. Progestogen-only hormonal contraception associated with the inhibition of ovulation; oral, intravaginal, transdermal.
   3. Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
   4. Male or female condom with or without spermicide
   5. Cap, diaphragm or sponge with spermicide
   6. Intrauterine device
   7. Intrauterine hormone-releasing system
   8. Bilateral tubal occlusion
   9. Vasectomised partner (where this was the subject's sole sexual partner and where the vasectomised partner had received medical assessment of the surgical success)
   10. Sexual abstinence (where the subject was willing to refrain from heterosexual intercourse during the entire period of the investigation in line with their preferred and usual lifestyle)

   Females who were considered to be of child-bearing potential were those who were fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause (Clinical Trials Facilitation Group, 2014).
8. Those who suffered from allergies or sensitivities to the raw material of the insoles (as detailed in the Investigator Brochure).
9. Those who had participated in another clinical investigation within the 3 months prior to enrolment into the run-in period.
10. Employee at the investigational site, or a partner or first degree relative of the Investigator or member of the investigation team at the site.
11. Those, in the opinion of the Investigator, who were not deemed suitable or were unable to comply fully with the investigation requirements, for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress. Assessed though the change in pain, measured by the Brief Pain Inventory questionnaire score. (For each of the four orthotic insoles separately.) | Time frame is dependent on working pattern Days 0-5 compared to Days 44-47 and Days 0-3 compared to Days 27-30
  The average change from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain) when compared to the first three days of the last working episode.
  To account for differences in subjects working patterns a definition was created, a valid working episode was considered to be two non-working days followed by at least three and up to five working days. (this definition was used for all outcomes)
  The baseline was defined as the first three consecutive working days of baseline working episode (Days 0-3). The first three days of the last working episode could occur from Days 27-30 for subjects that worked 3 consecutive working days up to Days 44-47 for subjects that worked five consecutive working days
  For each of the four orthotic insoles separately.

SECONDARY OUTCOMES:
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress over the first three days of each working episode. Assessed though change in pain, measured by the BPI. (For each of the four orthotic insoles) | Days 0-5 compared to Days 23-26, Days 30-33, Days 37-40, Days 0-3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 consecutive working days
  The average change from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), during the first three consecutive working days of each working episode (WE) of the treatment period
  The baseline WE was defined as the first three consecutive working days of (Days 0-3):
  1. st WE- the first three days could occur from Days 12-15 for subjects that worked 3 consecutive working days up to Days 23-26 for subjects that worked five consecutive working days
  2. nd WE- the first three days could occur from Days 17-20 for subjects that worked 3 consecutive working days up to Days 30-33 for subjects that worked five consecutive working days
  3. rd WE- the first three days could occur from Days 22-25 for subjects that worked 3 consecutive working days up to Days 37-40 for subjects that worked five consecutive working days
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress over each working episode. Assessed though change in pain, measured by the BPI questionnaire.(For each of the four orthotic insoles) | Days 0-5 compared to Day 23-28, Day 30-35, Day 37-42, Day 44-49 for subjects that worked five consecutive working days, Days 0-3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 consecutive working days
  The change from baseline in the composite score of the worse, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), completed at the end of each working episode (WE) of the treatment period.
  The baseline WE was defined as Days 0-3 or Days 0-5 depending on the working pattern of the subjects:
  1. st WE- the last working day could occur on Day 12-15 for subjects that worked 3 consecutive working days (CWD) up to Days 23-28 for subjects that worked 5 CWD
  2. nd WE- the last working day could occur on Day 17-20 for subjects that worked 3 CWD up to Day 30-35 for subjects that worked 5 CWD
  3. rd WE- the last working day of the 3rd working episode could occur from Day 22-25 for subjects that worked 3 CWD up to Day 37-42 for subjects that worked 5 CWD
  4. th WE- the last working day could occur from Day 27-30 for subjects that worked 3 CWD up to Day 44-49 for subjects that worked 5 CWD
Proportion of subjects who achieve a change of ≥1 unit from baseline Assessed though the change in pain, measured by the Brief Pain Inventory questionnaire score. (For each of the four orthotic insoles separately.) | Days 0-5 compared to Days 44-47 for subjects that worked 5 consecutive working days, Days 0-3 compared to Days 27-30 for subjects that worked 3 consecutive working days
  The overall proportion of subjects who achieve a change of ≥1 unit from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), during the first three consecutive working days of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  To account for differences in subjects working patterns a definition was created, a valid working episode was considered to be two non-working days followed by at least three and up to five working days .
  The baseline was defined as the first three consecutive working days of baseline working episode (Days 0-3). The first three days of the last working episode could occur from Days 27-30 for subjects that worked 3 consecutive working days up to Days 44-47 for subjects that worked five consecutive working days
Subject impression of change in pain (Visual Analogue Scale) (For each of the four orthotic insoles separately.) | Day 6 and Day 15 (Visit 1) compared to Day 31 and Day 50 depending on the subjects working pattern.
  Subjects' rating of overall improvement in pain since pre-treatment, completed at the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  Scored on a scale of -3 to +3 with 0 indicating no change in pain, a positive number indicating an improvement and negative indicating an increase in the pain
Investigator impression of change in subjects' pain (Visual Analogue Scale) (For each of the four orthotic insoles separately.) | Day 6 and Day 15 (Visit 1) compared to Day 31 and Day 50 depending on the subjects working pattern.
  Investigator's rating of the subjects' overall improvement in pain since pre-treatment, completed following the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  Scored on a scale of -3 to +3 with 0 indicating no change in pain, a positive number indicating an improvement and negative indicating an increase in the pain
Change in quality of life, associated with improvement pain as assessed by the Brief Pain Inventory questionnaire. (For each of the four orthotic insoles separately.) | Day 5 compared to Day 23-28, Day 30-35, Days 37-42 Day 44-49 for subjects that worked 5 CWD or Day 3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 CWD
  The change from baseline in quality of life, associated with overall improvement in pain in the primary area of pain, assessed by the Brief Pain Inventory pain (BPI) interference scores (Question 9; composite (average) score), completed at the end of each working episode (WE) of the treatment period.
  The baseline WE was defined as Day 3 or Days 5 depending on the working pattern:
  1. st WE- occurred from Day 12-15 for subjects that worked 3 consecutive working days (CWD) up to Day 23-28 for subjects that worked 5 CWD
  2. nd working episode- occurred from Day 17-20 for subjects that worked 3 CWD up to Day 30-35 for subjects that worked 5 CDW
  3. rd working episode- occurred from Day 22-25 for subjects that worked 3 CWD up to Day 37-42 for subjects that worked five consecutive working days
  4. th working episode- occurred from Day 27-30 for subjects that worked 3 CWD up to Day 44-49 for subjects that worked 5 CWD The BPI question is a scale of 0-10 with the lower number indicating less pain
Change in quality of life, associated with improvement in pain as assessed by the EQ-5D-5L (questionaire) (For each of the four orthotic insoles separately.) | Day 3 up to 5 compared to Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Change from baseline in quality of life, associated with overall improvement in pain in the primary area of pain, assessed by the EQ-5D-5L, completed at the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  The baseline was defined as the first three up to five consecutive working days of baseline working episode therefore in the context of this endpoint the baseline assessment would occur on Day 3 or Days 5 depending on the working pattern of the subjects. Compared to the responses at the end of last working episode which could occur from Day 30 for subjects that worked 3 consecutive working days up to Day 49 for subjects that worked five consecutive working days.
  The EuroQol-5 dimension-5 Level (EQ-5D-5L), is made up of 5 questions scored 1 to 5 from these questions an index is created with a range between zero and 1 with a zero being death and 1 being perfect quality of life.
Change in work productivity and activity as assessed by the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (For each of the four orthotic insoles separately.) | Quality of life on Day 3 up to 5 compared to Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Change from baseline in work productivity and activity, assessed by the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP), completed at the end of last working episode of the treatment period. For each of the four orthotic insoles separately.
  The baseline was defined as the first 3 up to 5 consecutive working days (CWD) of baseline working episode therefore in the context of this endpoint the baseline assessment would occur on Day 3 or Days 5 depending on the working pattern of the subjects. Compared to the responses at the end of last working episode which could occur from Day 30 for subjects that worked 3 CWD up to Day 49 for subjects that worked 5 CWD.
  The WPAI:SHP six questions on the subjects productivity and activity Impairment. Questions comprised of information on employment, including hours at work, hours missed from work and reasons for work missed. As well as the effect that pain had on their daily activities.
Subject impression of change in their work productivity and activity. (Visual Analogue Scale) (For each of the four orthotic insoles separately.) | Quality of life improvement assessed on Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Subjects' rating of overall improvement in their quality of life and work productivity and activity since pre-treatment, completed at the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  The last working day is therefore different for each subjects working pattern this could occur from Day 30 for subjects that worked 3 consecutive working days (CWD) up to Day 49 for subjects that worked 5 CWD.
  This assessment was scored on a scale of -3 to +3 with 0 indicating no change, a positive number indicating an improvement and negative indicating an increase in quality of life
Investigator impression of change in quality of life (Visual Analogue Scale) (For each of the four orthotic insoles separately.) | Quality of life improvement assessed on Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Investigator's rating of the subjects' overall improvement in their quality of life since pre-treatment, following the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  The last working day is therefore different for each subjects working pattern this could occur from Day 30 for subjects that worked 3 consecutive working days up to Day 49 for subjects that worked five consecutive working days.
  This assessment was scored on a scale of -3 to +3 with 0 indicating no change in quality of life, a positive number indicating an improvement and negative indicating an increase in quality of life
Safety and tolerability of the device (For each of the four orthotic insoles separately.) | through to study completion, from point of informed consent (Day 1) up to Visit 3 (Day 50)
  Overall proportion of subjects with AEs and adverse device effects (ADEs), i.e. the occurrence of one or more AEs/ADEs per subject. For each of the four orthotic insoles separately.

OTHER OUTCOMES:
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress during the first three days of the break-in working episode. As assessed by the change in BPI questionnaire. (For each of the four orthotic insoles) | Average pain on Days 0-3 compared to Days 7-10 for subjects that worked three consecutive working days, Average pain on Days 0-5 compared to Days 9-14 for subjects that worked five consecutive working days
  The average change from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), during the first three consecutive working days of the working episode (WE)of the breaking-in period.
  The baseline WE first 3 up to 5 consecutive working days (CWD) of baseline working episode therefore in the context of this endpoint the baseline assessment is an average of the responses Day 0-3 or Days 0-5 depending on the working pattern of the subjects.
  The break- in period was defined as the first working episode where the subject was provided with the device, it started with at least one non-working and included three up to five consecutive working days. For this endpoint the first three days would take place over Day 7-10.
  The average pain during the break-in period was compared to the baseline.
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress during the break-in working episode. As assessed by the change in the BPI score. (For each of the four orthotic insoles separately) | Average pain on Days 3 was compared that on Day 10 for subjects that worked three consecutive working days, Average pain on Days 5 compared to Day 14 for subjects that worked five consecutive working days.
  The change from baseline in the composite score of the worse, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), completed at the end of the working episode of the breaking-in period. For each of the four orthotic insoles separately.
  The baseline WE defined as the first 3 up to 5 consecutive working days (CWD) of baseline working episode therefore the baseline assessment would occur on Day 3 or Days 5 depending on the working pattern of the subjects.
  The break- in period was defined as the first working episode where the subject was provided with the device, at least one non-working and included three up to five CWD. For this endpoint the end of the working episode would occur on Day 10 or Day 14 depending on the working pattern of the subjects.
  The average pain at the end of the break-in period was compared to the baseline.
Change in quality of life, associated with improvement pain as assessed by the Brief Pain Inventory questionnaire following the break-in period (For each of the four orthotic insoles separately) | Day 5 compared to Day 23-28, Day 30-35, Days 37-42, Day 44-49 for subjects that worked five CWD or Day 3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 CWD
  The change from baseline in quality of life, associated with overall improvement in pain in the primary area of pain, assessed by the Brief Pain Inventory (BPI) pain interference scores (Question 9; composite (average) score), completed at the end of the working episode of the breaking-in period. For each of the four orthotic insoles separately.
  The baseline WE occurred on Day 3 or Days 5 depending on the working pattern:
  1. WE- occurred from Day 12-15 for subjects that worked 3 consecutive working days (CWD) up to Day 23-28 for subjects that worked 5 CWD
  2. WE- occurred from Day 17-20 for subjects that worked 3 CWD up to Day 30-35 for subjects that worked 5 CWD
  3. WE- occurred from Day 22-25 for subjects that worked 3 CWD up to Day 37-42 for subjects that worked 5 CWD
  4. WE- occurred from Day 27-30 for subjects that worked 3 CWD up to Day 44-49 for subjects that worked 5 CWD The BPI questions is on a scale of 0-10 with the lower number indicating less pain.
Subject perceived improvement of symptoms (questionnaire) (For each of the four orthotic insoles separately) | Days 11-21 of the full-use period for subjects that worked 3 consecutive working days. Days 22-32 of the full-use period for subjects that worked 5 consecutive working days.
  Improvement of symptoms as a result of wearing the insoles, recorded through a Subject Perceived Questions, daily for the first ten days of the treatment period. For each of the four orthotic insoles separately.
  This assessment was scored on five statements with the subject selecting the most appropriate statement with statement 1 being no change and statement 5 being completely better.
Subjects impressions of comfort and impact of insoles (questionnaire) (For each of the four orthotic insoles separately) | Daily though out the treatment period. Day 11 to Day 30 of the full-use period for subjects that worked 3 consecutive working days. Day 21 to 49 for subjects that worked 5 consecutive working days.
  Comfort of the insole and impact on daily activity, recorded through Subject Perceived Questions on a daily basis throughout the treatment period. For each of the four orthotic insoles separately.
  This assessment was scored on a scale of 0 to 10 with 0 being very uncomfortable and 10 very comfortable.
Subjects impressions tolerability (Visual Analogue Scale) (For each of the four orthotic insoles separately) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days.
  Subject impression of tolerability, as assessed through comfort, irritation and ADEs, completed at the end of the last working episode of the treatment period.
  This assessment was scored on a scale of -3 to +3 with 0 indicating no change, a positive number indicating well tolerated and negative indicating an not well tolerated.
Subject experience and satisfaction of insoles (Visual Analogue Scale) | Daily though out the treatment period. Day 11 to Day 30 of the full-use period for subjects that worked 3 consecutive working days. Day 21 to 49 for subjects that worked 5 consecutive working days.
  Overall subject experience and satisfaction completed at the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  Experience and satisfaction assessed as separately as two questions and scored on a scale of -3 to +3 with 0 indicating no change, a positive number indicating an improvement and negative number indicating a negative experience/ satisfaction.
Investigator impression of tolerability (Visual Analogue Scale) (For each of the four orthotic insoles separately) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days
  Overall subject experience and satisfaction, completed at the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  Experience and satisfaction assessed as separately as two questions and scored on a scale of -3 to +3 with 0 indicating no change, a positive number indicating an improvement and negative number indicating an negative experience/ satisfaction.
Investigator global impression of tolerability (Statement) (For each of the four orthotic insoles separately) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days
  Investigator global impression of tolerability, as assessed through comfort, irritation and ADEs across the investigation, completed following the end of the last working episode of the treatment period for the last subject. For each of the four orthotic insoles separately.
  Statement from the Investigator included within the Clinical Investigation Report
Subjects impressions (questionnaire) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days
  End of study Subject Perceived Questions, completed on the day of Visit 3. For each of the four orthotic insoles separately.
  Subjects answered questions with each question having five levels of agreement (strongly disagree to strongly agree), the subjects selected the most appropriate statement.
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress. Assessed though the change in pain, measured by the Brief Pain Inventory questionnaire. (analysed for all insoles collectively) | Time frame is dependent on working pattern Days 0-5 compared to Days 44-47 and Days 0-3 compared to Days 27-30
  The average change from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), during the first three consecutive working days of the last working episode of the treatment period.
  To account for differences in subjects working patterns a definition was created, a valid working episode was considered to be two non-working days followed by at least three and up to five working days .
  The baseline was defined as the first three consecutive working days of baseline working episode (Days 0-3). The first three days of the last working episode could occur from Days 27-30 for subjects that worked 3 consecutive working days up to Days 44-47 for subjects that worked five consecutive working days
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress over the first three days of each working episode. Assessed change in pain, measured by the BPI questionnaire. (analysed for all insoles) | Days 0-5 compared to Days 23-26, Days 30-33, Days 37-40, Days 0-3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 consecutive working days
  The average change from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), during the first three consecutive working days of each working episode (WE) of the treatment period
  The baseline WE was defined as the first three consecutive working days of (Days 0-3):
  1. st WE- the first three days could occur from Days 12-15 for subjects that worked 3 consecutive working days up to Days 23-26 for subjects that worked five consecutive working days
  2. nd WE- the first three days could occur from Days 17-20 for subjects that worked 3 consecutive working days up to Days 30-33 for subjects that worked five consecutive working days
  3. rd WE- the first three days could occur from Days 22-25 for subjects that worked 3 consecutive working days up to Days 37-40 for subjects that worked five consecutive working days
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress over each working episode. Assessed though the change in pain, measured by the BPI questionnaire.(analysed for all insoles collectively) | Days 0-5 compared to Day 23-28, Day 30-35, Day 37-42, Day 44-49 for subjects that worked five consecutive working days, Days 0-3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 consecutive working days
  The change from baseline in the composite score of the worse, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), completed at the end of each working episode (WE) of the treatment period.
  The baseline WE was defined as Days 0-3 or Days 0-5 depending on the working pattern of the subjects:
  1. WE- the last working day could occur on Day 12-15 for subjects that worked 3 consecutive working days (CWD) up to Days 23-28 for subjects that worked 5 CWD
  2. WE- the last working day could occur on Day 17-20 for subjects that worked 3 CWD up to Day 30-35 for subjects that worked 5 CWD
  3. WE- the last working day of the 3rd working episode could occur from Day 22-25 for subjects that worked 3 CWD up to Day 37-42 for subjects that worked 5 CWD
  4. WE- the last working day could occur from Day 27-30 for subjects that worked 3 CWD up to Day 44-49 for subjects that worked 5 CWD
Proportion of subjects who achieve a change of ≥1 unit from baseline.Assessed though the change in pain, measured by the Brief Pain Inventory questionnaire. (analysed for all insoles collectively) | Days 0-5 compared to Days 44-47 for subjects that worked 5 consecutive working days, Days 0-3 compared to Days 27-30 for subjects that worked 3 consecutive working days
  The overall proportion of subjects who achieve a change of ≥1 unit from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), during the first three consecutive working days of the last working episode of the treatment period.
  To account for differences in subjects working patterns a definition was created, a valid working episode was considered to be two non-working days followed by at least three and up to five working days .
  The baseline was defined as the first three consecutive working days of baseline working episode (Days 0-3). The first three days of the last working episode could occur from Days 27-30 for subjects that worked 3 consecutive working days up to Days 44-47 for subjects that worked five consecutive working days
Subject impression of change in pain (Visual Analogue Scale) (analysed for all insoles collectively) | Day 6 and Day 15 (Visit 1) compared to Day 31 and Day 50 depending on the subjects working pattern.
  Subjects' rating of overall improvement in pain since pre-treatment, completed at the end of the last working episode of the treatment period.
  Analysed for all insoles collectively.
  Scored on a scale of -3 to +3 with 0 indicating no change in pain, a positive number indicating an improvement and negative indicating an increase in the pain
Investigator impression of change in subjects' pain (Visual Analogue Scale) (analysed for all insoles collectively) | Day 6 and Day 15 (Visit 1) compared to Day 31 and Day 50 depending on the subjects working pattern.
  Investigator's rating of the subjects' overall improvement in pain since pre-treatment, completed following the end of the last working episode of the treatment period.
  Scored on a scale of -3 to +3 with 0 indicating no change in pain, a positive number indicating an improvement and negative indicating an increase in the pain
  Analysed for all insoles collectively.
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress during the first three days of the break-in working episode. Assessed change in pain, measured by the BPI questionnaire. (analysed for all insoles) | Average pain on Days 0-3 compared to Days 7-10 for subjects that worked three consecutive working days, Average pain on Days 0-5 compared to Days 9-14 for subjects that worked five consecutive working days
  The average change from baseline in the daily composite score of the worst, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), during the first three consecutive working days of the working episode (WE)of the breaking-in period.
  The baseline WE first 3 up to 5 consecutive working days (CWD) of baseline working episode therefore in the context of this endpoint the baseline assessment is an average of the responses Day 0-3 or Days 0-5 depending on the working pattern of the subjects.
  The break- in period was defined as the first working episode where the subject was provided with the device, it started with at least one non-working and included three up to five consecutive working days. For this endpoint the first three days would take place over Day 7-10.
  The average pain during the break-in period was compared to the baseline.
Evaluation of the pain relief caused by orthotic insoles on pain associated with musculoskeletal stress during the break-in working episode Assessed though the change in pain, measured by the BPI questionnaire.(analysed for all insoles collectively) | Average pain on Days 3 was compared that on Day 10 for subjects that worked three consecutive working days, Average pain on Days 5 compared to Day 14 for subjects that worked five consecutive working days.
  The change from baseline in the composite score of the worse, least, average and current pain, as measured by Questions 3-6 of the Brief Pain Inventory (BPI, scored on a scale of 0-10 with the lower number indicating less pain), completed at the end of the working episode of the breaking-in period. For each of the four orthotic insoles separately.
  The baseline WE defined as the first 3 up to 5 consecutive working days (CWD) of baseline working episode therefore the baseline assessment would occur on Day 3 or Days 5 depending on the working pattern of the subjects.
  The break- in period was defined as the first working episode where the subject was provided with the device, at least one non-working and included three up to five CWD. For this endpoint the end of the working episode would occur on Day 10 or Day 14 depending on the working pattern of the subjects.
  The average pain at the end of the break-in period was compared to the baseline.
Change in quality of life, associated with improvement pain as assessed by the Brief Pain Inventory questionnaire (analysed for all insoles collectively) | Day 5 compared to Day 23-28, Day 30-35, Days 37-42 Day 44-49 for subjects that worked 5 CWD or Day 3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 CWD
  The change from baseline in quality of life, associated with overall improvement in pain in the primary area of pain, assessed by the Brief Pain Inventory pain (BPI) interference scores (Question 9; composite (average) score), completed at the end of each working episode (WE) of the treatment period.
  The baseline WE was defined as Day 3 or Days 5 depending on the working pattern:
  1. st WE- occurred from Day 12-15 for subjects that worked 3 consecutive working days (CWD) up to Day 23-28 for subjects that worked 5 CWD
  2. nd working episode- occurred from Day 17-20 for subjects that worked 3 CWD up to Day 30-35 for subjects that worked 5 CDW
  3. rd working episode- occurred from Day 22-25 for subjects that worked 3 CWD up to Day 37-42 for subjects that worked five consecutive working days
  4. th working episode- occurred from Day 27-30 for subjects that worked 3 CWD up to Day 44-49 for subjects that worked 5 CWD The BPI question is a scale of 0-10 with the lower number indicating less pain.
Change in quality of life, associated with improvement in pain as assessed by the EQ-5D-5L questionnaire (analysed for all insoles collectively) | Day 3 up to 5 compared to Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Change from baseline in quality of life, associated with overall improvement in pain in the primary area of pain, assessed by the EQ-5D-5L, completed at the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  The baseline was defined as the first three up to five consecutive working days of baseline working episode therefore in the context of this endpoint the baseline assessment would occur on Day 3 or Days 5 depending on the working pattern of the subjects. Compared to the responses at the end of last working episode which could occur from Day 30 for subjects that worked 3 consecutive working days up to Day 49 for subjects that worked five consecutive working days.
  The EuroQol- 5 dimension - 5 level (EQ-5D-5L), is made up of 5 questions scored 1 to 5 from these questions an index is created with a range between zero and 1 with a zero being death and 1 being perfect quality of life.
Change in work productivity and activity as assessed by the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (analysed for all insoles collectively) | Quality of life on Day 3 up to 5 compared to Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Change from baseline in work productivity and activity, assessed by the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP), completed at the end of last working episode of the treatment period. For each of the four orthotic insoles separately.
  The baseline was defined as the first 3 up to 5 consecutive working days (CWD) of baseline working episode therefore in the context of this endpoint the baseline assessment would occur on Day 3 or Days 5 depending on the working pattern of the subjects. Compared to the responses at the end of last working episode which could occur from Day 30 for subjects that worked 3 CWD up to Day 49 for subjects that worked 5 CWD.
  The WPAI:SHP six questions on the subjects productivity and activity Impairment. Questions comprised of information on employment, including hours at work, hours missed from work and reasons for work missed. As well as the effect that pain had on their daily activities..
Subject impression of change in their work productivity and activity. (Visual Analogue Scale) (analysed for all insoles collectively) | Quality of life improvement assessed on Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Subjects' rating of overall improvement in their quality of life and work productivity and activity since pre-treatment, completed at the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  The last working day is different for each subject working pattern this could occur from Day 30 for subjects that worked 3 consecutive working days (CWD) up to Day 49 for subjects that worked 5 CWD.
  This assessment was scored on a scale of -3 to +3 with 0 indicating no change, a positive number indicating an improvement and negative indicating an increase in quality of life
Investigator impression of change in quality of life (Visual Analogue Scale) (analysed for all insoles collectively) | Quality of life improvement assessed on Day 49 for subjects that worked five consecutive working days or Day 30 for subjects that worked 3 consecutive working days
  Investigator's rating of the subjects' overall improvement in their quality of life since pre-treatment, following the end of the last working episode of the treatment period. For each of the four orthotic insoles separately.
  The last working day is therefore different for each subjects working pattern this could occur from Day 30 for subjects that worked 3 consecutive working days up to Day 49 for subjects that worked five consecutive working days.
  This assessment was scored on a scale of -3 to +3 with 0 indicating no change in quality of life, a positive number indicating an improvement and negative indicating an increase in quality of life
Safety and tolerability of the device (analysed for all insoles collectively) | through study completion, from point of informed consent (Day 1) up to Visit 3 (Day 50)
  Overall proportion of subjects with AEs and adverse device effects (ADEs), i.e. the occurrence of one or more AEs/ADEs per subject.
  Analysed for all insoles collectively.
Change in quality of life, associated with improvement pain as assessed by the Brief Pain Inventory following the break-in period (analysed for all insoles collectively) | Day 5 compared to Day 23-28, Day 30-35, Days 37-42, Day 44-49 for subjects that worked five CWD or Day 3 compared to Day 12-15, Day 17-20, Day 22-25, Day 27-30 for subjects that worked 3 CWD
  The change from baseline in quality of life, associated with overall improvement in pain in the primary area of pain, assessed by the Brief Pain Inventory (BPI) pain interference scores (Question 9; composite (average) score), completed at the end of the working episode of the breaking-in period. For each of the four orthotic insoles separately.
  The baseline WE occurred on Day 3 or Days 5 depending on the working pattern:
  1. WE- occurred from Day 12-15 for subjects that worked 3 consecutive working days (CWD) up to Day 23-28 for subjects that worked 5 CWD
  2. WE- occurred from Day 17-20 for subjects that worked 3 CWD up to Day 30-35 for subjects that worked 5 CWD
  3. WE- occurred from Day 22-25 for subjects that worked 3 CWD up to Day 37-42 for subjects that worked 5 CWD
  4. WE- occurred from Day 27-30 for subjects that worked 3 CWD up to Day 44-49 for subjects that worked 5 CWD The BPI questions is on a scale of 0-10 with the lower number indicating less pain.
Subject perceived improvement of symptoms (questionnaire) (analysed for all insoles collectively) | Days 11-21 of the full-use period for subjects that worked 3 consecutive working days. Days 22-32 of the full-use period for subjects that worked 5 consecutive working days.
  Improvement of symptoms as a result of wearing the insoles, recorded through a Subject Perceived Questions, daily for the first ten days of the treatment period. Analysed for all insoles collectively.
  This assessment was scored on five statements with the subject selecting the most appropriate statement with statement 1 being no change and statement 5 being completely better.
Subjects impressions of comfort and impact of insoles (questionnaire) (analysed for all insoles collectively) | Daily though out the treatment period. Day 11 to Day 30 of the full-use period for subjects that worked 3 consecutive working days. Day 21 to 49 for subjects that worked 5 consecutive working days.
  Comfort of the insole and impact on daily activity, recorded through Subject Perceived Questions on a daily basis throughout the treatment period. Analysed for all insoles collectively.
  This assessment was scored on a scale of 0 to 10 with 0 being very uncomfortable and 10 very comfortable.
Subjects impressions of tolerability (Visual Analogue Scale) (analysed for all insoles collectively) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days.
  Subject impression of tolerability, as assessed through comfort, irritation and ADEs, completed at the end of the last working episode of the treatment period. Analysed for all insoles collectively.
  This assessment was scored on a scale of -3 to +3 with 0 indicating no change, a positive number indicating well tolerated and negative indicating an not well tolerated.
Subjects experience and satisfaction of insoles (Visual Analogue Scale) (analysed for all insoles collectively) | Daily though out the treatment period. Day 11 to Day 30 of the full-use period for subjects that worked 3 consecutive working days. Day 21 to 49 for subjects that worked 5 consecutive working days.
  Overall subject experience and satisfaction, completed at the end of the last working episode of the treatment period.
  Analysed for all insoles collectively.
  Experience and satisfaction assessed as separately as two questions and scored on a scale of -3 to +3 with 0 indicating no change, a positive number indicating an improvement and negative number indicating an negative experience/ satisfaction.
Investigator impression of tolerability (Visual Analogue Scale) (analysed for all insoles collectively) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days
  Investigator impression of tolerability, as assessed through comfort, irritation and ADEs, completed following the end of the last working episode of the treatment period for each subject.
  Analysed for all insoles collectively.
  This assessment was scored on a scale of -3 to +3 with 0 indicating no change indifferent, a positive number indicating well tolerated and negative indicating not well tolerated
Investigator global impression of tolerability(Statement) (analysed for all insoles collectively) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days
  Investigator global impression of tolerability, as assessed through comfort, irritation and ADEs across the investigation, completed following the end of the last working episode of the treatment period for the last subject.
  Analysed for all insoles collectively.
  Statement from the Investigator included within the Clinical Investigation Report
Subjects impressions (Questionnaires) (analysed for all insoles collectively) | Day 31 for subjects that worked 3 consecutive working days. Day 50 for subjects that worked 5 consecutive working days
  End of study Subject Perceived Questions, completed on the day of Visit 3.
  Analysed for all insoles collectively.
  Subjects answered questions with each question having five levels of agreement (strongly disagree to strongly agree), the subjects selected the most appropriate statement.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Crawford, BSc (Hons), MBChB, Principal Investigator — Gordon.crawford@cpsresearch.co.uk
Locations (1):
- CPS Research, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida JS, Vanderlei FM, Pastre EC, Martins RA, Padovani CR, Filho GC. Comparison of Two Types of Insoles on Musculoskeletal Symptoms and Plantar Pressure Distribution in a Work Environment: A Randomized Clinical Trial. Clin Med Res. 2016 Jun;14(2):67-74. doi: 10.3121/cmr.2016.1301. Epub 2016 May 26. PMID 27231116
- [Background] Amer AO, Jarl GM, Hermansson LN. The effect of insoles on foot pain and daily activities. Prosthet Orthot Int. 2014 Dec;38(6):474-80. doi: 10.1177/0309364613512369. Epub 2013 Dec 13. PMID 24335153
- [Background] Basford JR, Smith MA. Shoe insoles in the workplace. Orthopedics. 1988 Feb;11(2):285-8. doi: 10.3928/0147-7447-19880201-08. PMID 2965809
- [Background] Bonanno DR, Landorf KB, Munteanu SE, Murley GS, Menz HB. Effectiveness of foot orthoses and shock-absorbing insoles for the prevention of injury: a systematic review and meta-analysis. Br J Sports Med. 2017 Jan;51(2):86-96. doi: 10.1136/bjsports-2016-096671. Epub 2016 Dec 5. PMID 27919918
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Gill TK, Menz HB, Landorf KB, Arnold JB, Taylor AW, Hill CL. Identification of Clusters of Foot Pain Location in a Community Sample. Arthritis Care Res (Hoboken). 2017 Dec;69(12):1903-1908. doi: 10.1002/acr.23212. Epub 2017 Nov 14. PMID 28229556
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Shabat S, Gefen T, Nyska M, Folman Y, Gepstein R. The effect of insoles on the incidence and severity of low back pain among workers whose job involves long-distance walking. Eur Spine J. 2005 Aug;14(6):546-50. doi: 10.1007/s00586-004-0824-z. Epub 2005 Jan 25. PMID 15668775
- [Background] Sobel E, Levitz SJ, Caselli MA, Christos PJ, Rosenblum J. The effect of customized insoles on the reduction of postwork discomfort. J Am Podiatr Med Assoc. 2001 Nov-Dec;91(10):515-20. doi: 10.7547/87507315-91-10-515. PMID 11734607
- [Background] Stanhope J. Brief Pain Inventory review. Occup Med (Lond). 2016 Aug;66(6):496-7. doi: 10.1093/occmed/kqw041. Epub 2016 Apr 11. No abstract available. PMID 27067913
- [Background] Stolt M, Suhonen R, Virolainen P, Leino-Kilpi H. Lower extremity musculoskeletal disorders in nurses: A narrative literature review. Scand J Public Health. 2016 Feb;44(1):106-15. doi: 10.1177/1403494815602989. Epub 2015 Sep 9. PMID 26355119
- [Background] Waters TR, Dick RB. Evidence of health risks associated with prolonged standing at work and intervention effectiveness. Rehabil Nurs. 2015 May-Jun;40(3):148-65. doi: 10.1002/rnj.166. Epub 2014 Jul 7. PMID 25041875